CLINICAL TRIAL: NCT07067996
Title: Erector Spinae Plane Block for Analgesia During ESWL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amr Abdelsabor, Resident, Anesthesia,Sugical Icu,Pain management Faculty of Medicine Sohag Univesity, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Soh-Med--25-6-8MS
Record Dates: First submitted 2025-07-06; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Renal Stone
MeSH Terms: conditions — Nephrolithiasis | interventions — Nalbuphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A : will receive Erector Spinae Plane Block in the prone position after URS. (Active Comparator): * Patients in the block group (Group A)will receive the ESPB in the prone position after URS. ESPB needle insertion sites will be tolerated to the location of the stone, between T7-T10 vertebra levels. With these adjustments, Following the marking of the thoracic vertebrae levels with a marker pen,
  * The intervention will be initiated when the transverse processes and costotransverse joints on the relevant level will be distinguished using a high frequency(10-15 MHZ) linear ultrasound probe. The needle will be inserted at a 30° angle to the skin in an in-plane and craniocaudal fashion
  * Proper placement will be confirmed with ultrasonography and then 20 mL of 0.25% bupivacaine solution&5 ml lidocaine 1% will be administered through the needle for intraoperative and postoperative anaglesia.
  Interventions: Procedure: erector spinae plane block
- group B : will receive nalbuphine (Active Comparator): •(Group B) patients will receive opioids ,nalbuphine( ,1 )mg/kg over 10 minutes then repeat the dose if needed &monitoring patients for respiratory depression
  Interventions: Drug: Nalbuphine

INTERVENTIONS:
Procedure: erector spinae plane block — erector spinae plane block will be given as intraoperive analgesia for patients undergoing Extracorporeal shock wave lithotripsy
  Arms: group A : will receive Erector Spinae Plane Block in the prone position after URS.
Drug: Nalbuphine — Nalbuphine will be given as intraopertive analgesia for patients undergoing Extracorporeal shock wave lithotripsy
  Arms: group B : will receive nalbuphine

SUMMARY:
this study aims to compare between efficacy of erector spinae plane block and conventional multimodal analgesia in Extracorporeal shock wave lithotripsy

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients undergoing ESWL with 2-3 cm renal stones
* patients between the ages of 21 and 60,
* both sexes,
* BMI ≥18≤30 kg/m²
* Able to give informed consent.
* Patients older than 18 years with American Society of Anesthesiologists Physical Status I or II and

Exclusion Criteria:

* Coagulopathy or on anticoagulants
* Infection at the ESPB injection site
* BMI ≥30 kg/m²
* Patient refusal.
* patients with advanced respiratory, renal, hepatic, neurological, or psychiatric disease, pregnant or nursing women.
* patients with a history of allergies to any study drugs

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
This study aims to evaluate the efficacy of Erector Spinae Plane Block analgesia for patients undergoing ESWL &compare between it and conventional multimodal Analgesia . | 6 hours postopertive
  postoperative pain by visual analog score from 0 to 10 (where 0 indicates no pain and 10 the worst possible pain

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Result] Karaaslan M, Olcucuoglu E, Kurtbeyoglu S, Tonyali S, Yilmaz M, Odabas O. Erector spinae plane block prior to extracorporeal shock wave lithotripsy decreases fluoroscopy time and promise a comfortable procedure for renal stones: A prospective randomized study. Actas Urol Esp (Engl Ed). 2023 Nov;47(9):566-572. doi: 10.1016/j.acuroe.2023.04.001. Epub 2023 Apr 20. English, Spanish. PMID 37084807
- [Result] Yayik AM, Ahiskalioglu A, Erguney OD, Oral Ahiskalioglu E, Alici H, Demirdogen SO, Adanur S. Analgesic efficacy of ultrasound-guided quadratus lumborum block during extracorporeal shock wave lithotripsy. Agri. 2020 Jan;32(1):44-47. doi: 10.5505/agri.2017.54036. PMID 32030700
- [Result] Alhashemi JA, Kaki AM. Dexmedetomidine in combination with morphine PCA provides superior analgesia for shockwave lithotripsy. Can J Anaesth. 2004 Apr;51(4):342-7. doi: 10.1007/BF03018237. PMID 15064262